CLINICAL TRIAL: NCT02946892
Title: Effect of Carvedilol on Exercise Performance in Fontan Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Principal Investigator, Ryan Butts, ASSOC PROFESSOR, PD-Cardiology, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 062016-101
Record Dates: First submitted 2016-09-23; First posted 2016-10-27 (Estimated); Results first posted 2021-01-22 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Single Ventricle; Fontan
MeSH Terms: conditions — Univentricular Heart | interventions — Carvedilol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Carvedilol (Experimental): Study participants will receive carvedilol for 12 weeks
  Interventions: Drug: Carvedilol
- Placebo (Experimental): Study participants will receive placebo (sugar pill) for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Carvedilol — Carvedilol will be given for 12 weeks and then an exercise test will be performed
  Other Names: Coreg
  Arms: Carvedilol
Drug: Placebo — Placebo will be given for 12 weeks and then an exercise test will be performed
  Other Names: Carvedilol Placebo
  Arms: Placebo

SUMMARY:
This study evaluates the effect of carvedilol in patients who have undergone a Fontan heart operation. All participants will receive carvedilol and placebo for 12 weeks. Exercise tests will be performed at the end of each 12 week period.

DETAILED DESCRIPTION:
Carvedilol is a well studied heart failure medication in adult heart failure that has been shown to improve outcomes. However, it has not been studied in patients who have had a Fontan heart operation. Study participants will receive either placebo or carvedilol for 12 weeks, at the end of the 12 weeks participants will perform an exercise test. Then study participants will receive treatment with placebo or carvedilol for 12 weeks (opposite of what participants go the first 12 weeks) and will again perform an exercise test.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent of parent(s) or legal guardian; informed consent or assent of subject as applicable.
2. Male or female children between the ages of 10 and 35 years with congenital heart disease that has been palliated with a Fontan circulation.
3. Ability of perform a maximal exercise test as defined by a respiratory exchange ratio (RER) greater than 1.0 at the time of maximal exercise

Exclusion Criteria:

1. The use of beta blockers within 2 months of randomization
2. Patients actively listed for transplantation at time of entry into the study or anticipated to undergo heart transplantation, interventional catheterization, or corrective cardiac surgery during the 7 months following entry into the study
3. Sustained or symptomatic ventricular dysrhythmias uncontrolled by drug therapy or the use of an implantable defibrillator, and/or significant cardiac conduction defects, e.g., 2nd degree or 3rd degree AV block, or sick sinus syndrome, unless a functioning pacemaker is in place
4. Uncorrected obstructive or severe regurgitant valve disease, nondilated cardiomyopathy, or significant systemic ventricular outflow obstruction
5. Known renovascular hypertension or evidence of pulmonary hypertension (pulmonary vascular resistance > 6 Wood units) unresponsive to vasodilator agents such as oxygen, nitroprusside, or nitric oxide
6. History or current clinical evidence of moderate-to-severe fixed obstructive pulmonary disease or severe reactive airway diseases (e.g., asthma) requiring hospitalization within the past 2 years or patient currently using long-term inhaled bronchodilators
7. Renal, hepatic, gastrointestinal, or biliary disorder that could impair absorption, metabolism or excretion of orally administered medication
8. Concurrent terminal illness or other severe disease (e.g., active neoplasm) or other significant laboratory value(s) which, in the opinion of the investigator, could preclude participation or survival
9. Endocrine disorders such as primary aldosteronism, pheochromocytoma, hyper- or hypothyroidism, insulin-dependent diabetes mellitus
10. Unwillingness or inability to cooperate, or for the parents or guardians to give consent, or for the child to give assent, or any condition of sufficient severity to impair cooperation in the study
11. Pregnancy or possible pregnancy at time of randomization, or female of child bearing potential who are lactating, or sexually active and not taking adequate contraceptive precautions (e.g., intrauterine device or oral contraceptives for 3 months prior to entry into the study)
12. Use of an investigational drug within 30 days of randomization, or within 5 half-lives of the investigational drug (the longer period will apply)
13. History of drug sensitivity or allergic reaction to alpha-blockers or ß-blockers
14. Use of any of the following medications within two weeks of randomization: MAO inhibitors, Calcium channel blockers, alpha blockers, beta blockers, disopyramide, flecainide, encainide, moricizine, propafenone, sotalol, or beta adrenergic agonists
15. Hospital admission for protein losing enteropathy or plastic bronchitis within 3 months of randomization
16. Active and/or chronic protein losing enteropathy or plastic bronchitis (on inhaled medication to control the plastic bronchitis).
17. Hypoalbuminemia defined as serum albumin <2.0g/dL
18. Renal dysfunction defined as serum creatinine >2.0mg/dL
19. Hepatic dysfunction defined as serum AST and/or ALT> 3 times upper limit of normal (approximately 120 IU/L however, will vary depending on age),
20. Significant anemia or polycythemia defined as hemoglobin >18gm/dL or hemoglobin <7gm/dL
21. Severely elevated serum BNP defined as BNP>300pg/ml

Ages: 10 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 26 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2020-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas Southwestern, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Butts R, Atz AM, BaezHernandez N, Sutcliffe D, Reisch J, Mahony L. Carvedilol Does Not Improve Exercise Performance in Fontan Patients: Results of a Crossover Trial. Pediatr Cardiol. 2021 Apr;42(4):934-941. doi: 10.1007/s00246-021-02565-6. Epub 2021 Feb 14. PMID 33585998

RESULTS

PARTICIPANT FLOW:
Groups:
- Carvedilol First, Then Placebo: Study participants will receive carvedilol for 12 weeks, washout for 6 weeks, then placebo for 12 weeks
- Placebo First, Then Carvedilol: Study participants will receive placebo (sugar pill) for 12 weeks, then washout for 6 weeks, then carvedilol for 12 weeks
Period: First Intervention (12 Weeks)
Arm/Group | Carvedilol First, Then Placebo | Placebo First, Then Carvedilol
Started | 11 | 15
Completed | 11 | 14
Not Completed | 0 | 1
Period: Washout (6 Weeks)
Arm/Group | Carvedilol First, Then Placebo | Placebo First, Then Carvedilol
Started | 11 | 14
Completed | 9 | 14
Not Completed | 2 | 0
Period: Second Intervention
Arm/Group | Carvedilol First, Then Placebo | Placebo First, Then Carvedilol
Started | 9 | 14
Completed | 9 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Since All Participants Would Be Randomized to Both Interventions, all Patients were Analyzed
Arm/Group | All Study Participants
Number analyzed (Participants) | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.9 (2.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 17
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-Caucasian | 5
  Caucasian | 18
Region of Enrollment [Number; unit: participants]
  United States | 23

OUTCOME MEASURES:

1. Primary Outcome: Change in Peak Oxygen Uptake From Baseline Peak Oxygen Uptake
Description: during exercise test on week 12 and week 30
Time Frame: on week 12 and week 30 of the study
Measure: Mean (Standard Deviation); unit: ml/kg/min
Arm/Group | Carvedilol | Placebo
Number analyzed (Participants) | 23 | 23
ml/kg/min | -2.01 (3.57) | -1.01 (3.36)

2. Secondary Outcome: Change in Peak Heart Rate
Description: during exercise test on week 12 and week 30
Time Frame: on week 12 and week 30 of the study
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Carvedilol | Placebo
Number analyzed (Participants) | 23 | 23
beats per minute | -32.3 (24.2) | 1.9 (12.6)

3. Secondary Outcome: Change in Oxygen Uptake at Anaerobic Threshold
Description: during exercise test on week 12 and week 30
Time Frame: on week 12 and week 30 of the study
Measure: Mean (Standard Deviation); unit: ml/kg/min
Arm/Group | Carvedilol | Placebo
Number analyzed (Participants) | 23 | 23
ml/kg/min | -1.02 (3.75) | -1.78 (4.55)

ADVERSE EVENTS:
Time Frame: 36 weeks
Description: AE were classified as serious or non-serious also related to study drug or unrelated to study drug at the time of the study visit.
Arm/Group | Carvedilol | Placebo
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/24
Other Adverse Events (participants affected / at risk) | 4/25 | 0/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Carvedilol (N=25) | Placebo (N=24)
Bradycardia (Cardiac disorders) | 4 (4) | 0 (0) — Low Heart Rate

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-02): https://cdn.clinicaltrials.gov/large-docs/92/NCT02946892/Prot_SAP_000.pdf